CLINICAL TRIAL: NCT00383799
Title: Comparison of Intravenous Amiodarone Versus Intravenous Procainamide for the Acute Treatment of Regular and Haemodynamically Well Tolerated Wide QRS Tachycardia (Probably of Ventricular Origen). The PROCAMIO Multicenter Study
Brief Title: Iv Amiodarone Versus Iv Procainamide to Treat Haemodynamically Well Tolerated Ventricular Tachycardia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Steering Committee decision after inclusion of 74 patients after 6 years and very slow inclusion rate
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001505-25
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Ventricular Tachycardia; Wide QRS Tachycardia
Keywords: Ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Amiodarone; Procainamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): IV procainamide (single dose: 10 mg/kg over 20 min)
  Interventions: Drug: iv Procainamide
- Group 2 (Active Comparator): IV Amiodarone (single dose: 5 mg/kg over 20 min)
  Interventions: Drug: iv Amiodarone

INTERVENTIONS:
Drug: iv Amiodarone
  Arms: Group 2
Drug: iv Procainamide
  Arms: Group 1

SUMMARY:
The purpose of this study is to determine whether intravenous amiodarone has less cardiac significant adverse events compared to intravenous procainamide in the acute treatment of haemodynamically well tolerated wide QRS tachycardia, the majority of them of probably ventricular origen.

DETAILED DESCRIPTION:
Multicenter, prospective and randomized study in phase IV. A total of 302 patients will be included in the study within 40-50 institutions in Spain. Patients with regular and monomorphic tachycardia ≥ 120 bpm, QRS ≥ 120 ms and haemodynamically well tolerated will be randomized to receive iv amiodarone (single dosage: 5 mg/kg in 20 minutes) vs iv procainamide (single dosage: 10 mg/kg in 20 minutes). The study period will be 40 minutes from infusion initiation. Study variables include the presence of clinically cardiac significant adverse events: hypotension, syncope, heart failure, symptomatic sinus bradycardia, AV block, proarrhythmia and tachycardia acceleration (<20 lpm)and death. Total observation period will be 24 hours after the end of the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable tachycardia ≥120 lpm, QRS ≥120 ms and haemodynamically well tolerated defined as: 1)Systolic blood pressure ≥90 mmHg, 2) absence of dyspnea at rest, 3)absence of peripheric hypoperfusion signs and 4)no severe angina.
* Age > 18 years
* Written inform consent obtained

Exclusion Criteria:

* Treatment with iv amiodarone or iv procainamide during the previous 24 hours
* QRS tachycardia <120 ms
* Patients with QRS ≥120 ms tachycardia with haemodynamic compromise that requires urgent cardioversion for termination
* Irregular tachycardia
* Tachycardia that is considered as supraventricular due to physician criteria (adenosine and/or vagal manoeuvres response)
* Patient that do not want to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To compare clinically significant cardiac adverse events occurring within 40 minutes from treatment initiation | 40 minutes

SECONDARY OUTCOMES:
To compare efficacy of both therapies in relation to episode termination | 40 minuutes
To compare the rate of total adverse events, cardiac and non cardiac, occurring during an observation period of 24 hours after treatment was applied | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Almendral, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón. Madrid. Spain; Fernando Arribas, MD, Study Director — Hospital General Universitario 12 de Octubre. Madrid. Spain; Rafael Peinado, MD, Study Director — Hospital General Universitario La Paz. Madrid. Spain; Alfonso Martín, MD, Study Director — Hospital de Móstoles. Madrid. Spain; Carmen del Arco, MD, Study Director — Hospital de la Princesa. Madrid. Spain; Dolores Vigil, MD, Study Director — Hospital general Universitario Gregorio Marañón. Madrid. Spain; Mercedes Ortiz, PhD, Study Director — Hospital General Universitario Gregorio Marañón. Madrid. Spain; Blanca Coll-Vinent, MD, Study Director — Hospital Clinic. Barcelona. Spain
Locations (29):
- Spain (29):
  - Hospital El Escorial, El Escorial, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Santa María del Rosell, Cartagena, Murcia
  - Fundación Hospitalaria de Cieza, Cieza, Murcia
  - Hospital Los Arcos, San Javier, Murcia
  - Hospital General, Alicante
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital San Cecilio, Granada
  - Hospital Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital de Móstoles, Madrid
  - Hospital General Universitario La Paz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de Son Dureta, Palma de Mallorca
  - Hospital de Son Llatzer, Palma de Mallorca
  - Hospital de Donostia, San Sebastián
  - Hospital de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hopital Clínico Universitario, Valencia
  - Hospital Río Hortega, Valladolid

REFERENCES:
- [Background] Guidelines 2000 for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Part 6: advanced cardiovascular life support: section 5: pharmacology I: agents for arrhythmias. The American Heart Association in collaboration with the International Liaison Committee on Resuscitation. Circulation. 2000 Aug 22;102(8 Suppl):I112-28. No abstract available. PMID 10966669
- [Background] ECC Committee, Subcommittees and Task Forces of the American Heart Association. 2005 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2005 Dec 13;112(24 Suppl):IV1-203. doi: 10.1161/CIRCULATIONAHA.105.166550. Epub 2005 Nov 28. No abstract available. PMID 16314375
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Blanc JJ, Budaj A, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (writing committee to develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Sep 5;114(10):e385-484. doi: 10.1161/CIRCULATIONAHA.106.178233. Epub 2006 Aug 25. No abstract available. PMID 16935995
- See also: Protocol home's page — https://operation.kikamedical.com/procamio